CLINICAL TRIAL: NCT05698446
Title: Comparison of Modified Broström Repair + Suture Tape and Anatomic Reconstruction for CLAI in Chronic Lateral Ankle Instability in Generalized Joint Laxity Cases: A Prospective Cohort Study
Brief Title: Comparison of MBR + Suture Tape, MBR, and Anatomic Reconstruction for CLAI in GJL Cases: A Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jiang Dong, Chief physician, Peking University Third Hospital
Other Study IDs: M2022514
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Ankle Sprains; Hypermobility Syndrome
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Open Modified Broström +Suture tape augmentation group: Patients who accept a modified Broström +Suture tape augmentation operation
  Interventions: Procedure: Modified Broström + Suture tape augmentation operation
- Anatomic reconstruction operation group: Patients who accept an anatomic reconstruction
  Interventions: Procedure: Anatomic reconstruction operation
- Open Modified Broström group: Patients who under went open Modified Broström-Gould surgery
  Interventions: Procedure: Open Modified Broström procedure

INTERVENTIONS:
Procedure: Modified Broström + Suture tape augmentation operation — Patients with CLAI and GJL will accept the Modified Broström + Suture tape augmentation operation
  Groups: Open Modified Broström +Suture tape augmentation group
Procedure: Anatomic reconstruction operation — Anatomic reconstruction operation
  Groups: Anatomic reconstruction operation group
Procedure: Open Modified Broström procedure — Open Modified Broström-Gould surgery
  Groups: Open Modified Broström group

SUMMARY:
GJL is a risk factor for postoperative recurrent instability following an MBR for CLAI. BPR with suture tape augmentation and anatomic reconstruction may provide more strength and stability. However, BPR with suture tape augmentation may lead to rejection of the suture tape, while anatomic reconstruction may be associated with more trauma. In addition, the outcomes between the BPR with suture tape augmentation and anatomic reconstruction were unknown.

DETAILED DESCRIPTION:
Generalized joint laxity (GJL) is a risk factor for postoperative recurrent instability following an open modified Broström repair (MBR) for chronic lateral ankle instability (CLAI). MBR with suture tape augmentation and anatomic reconstruction may provide more strength and stability. However, BPR with suture tape augmentation may lead to rejection of the suture tape, while anatomic reconstruction may be associated with more trauma. In addition, the outcomes between the BPR with suture tape augmentation and anatomic reconstruction were unknown.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lateral ankle pain and instability Beighton score ≥4 Age with 18 to 60 years

Exclusion Criteria:

* Patients with an acute or subacute ankle injury (within 3 months) Injury of the deltoid ligament Alignment of lower extremity greater than 5 degrees Fractures of the lower extremity Stage III or IV osteoarthritis Patients who refused to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patients who go to visit a doctor for persistent lateral ankle pain and instability over three months and invalid conservative treatment, with the age of 18- 60 years. If the Beighton score of the patient is ≥4 and the exclusion criteria are met, he or she is going to be advised to participate in this study.
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Karlsson-Peterson score | postoperative Karlsson score at 1 year
  This score is a primary scale for lateral ankle instability, with a maximum value of 100 and minimum value of 0. Larger Karlsson-Peterson score represents better ankle functional outcomes.
Karlsson-Peterson score | postoperative Karlsson score at 2 years
  This score is a primary scale for lateral ankle instability, with a maximum value of 100 and minimum value of 0. Larger Karlsson-Peterson score represents better ankle functional outcomes.

SECONDARY OUTCOMES:
Anterior displacement and talar tilt angle in stress radiography | postoperative radiographic measures at 2 years
  The outcomes are common indicators for evaluation the lateral stability of ankle

OTHER OUTCOMES:
Rate of re-injury | the rate of re-injury at 2 years
  After surgery, the rate of patients re-sprain

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The demographics data, Beighton score, primary and secondary outcomes would be available to other researchers

REFERENCES:
- [Background] Xu HX, Lee KB. Modified Brostrom Procedure for Chronic Lateral Ankle Instability in Patients With Generalized Joint Laxity. Am J Sports Med. 2016 Dec;44(12):3152-3157. doi: 10.1177/0363546516657816. Epub 2016 Aug 5. PMID 27496909
- [Background] Sacks HA, Prabhakar P, Wessel LE, Hettler J, Strickland SM, Potter HG, Fufa DT. Generalized Joint Laxity in Orthopaedic Patients: Clinical Manifestations, Radiographic Correlates, and Management. J Bone Joint Surg Am. 2019 Mar 20;101(6):558-566. doi: 10.2106/JBJS.18.00458. No abstract available. PMID 30893238
- [Background] Lan R, Piatt ET, Bolia IK, Haratian A, Hasan L, Peterson AB, Howard M, Korber S, Weber AE, Petrigliano FA, Tan EW. Suture Tape Augmentation in Lateral Ankle Ligament Surgery: Current Concepts Review. Foot Ankle Orthop. 2021 Oct 20;6(4):24730114211045978. doi: 10.1177/24730114211045978. eCollection 2021 Oct. PMID 35097476
- [Background] Michels F, Cordier G, Burssens A, Vereecke E, Guillo S. Endoscopic reconstruction of CFL and the ATFL with a gracilis graft: a cadaveric study. Knee Surg Sports Traumatol Arthrosc. 2016 Apr;24(4):1007-14. doi: 10.1007/s00167-015-3779-1. Epub 2015 Sep 26. PMID 26410096
- [Background] Cho BK, Park JK, Choi SM, SooHoo NF. A randomized comparison between lateral ligaments augmentation using suture-tape and modified Brostrom repair in young female patients with chronic ankle instability. Foot Ankle Surg. 2019 Apr;25(2):137-142. doi: 10.1016/j.fas.2017.09.008. Epub 2017 Oct 18. PMID 29409289